CLINICAL TRIAL: NCT01828489
Title: NOPHO-DBH AML 2012 Protocol. Research Study for Treatment of Children and Adolescents With Acute Myeloid Leukaemia 0-18 Years
Brief Title: Research Study for Treatment of Children and Adolescents With Acute Myeloid Leukaemia 0-18 Years
Acronym: AML2012
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NOPHO-DBH-AML2012; 2012-002934-35 (EudraCT Number)
Record Dates: First submitted 2013-04-06; First posted 2013-04-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Pediatric Acute Myeloblastic Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard arm MEC and ADxE (Active Comparator): Standard protocol arm with mitoxantrone in first course (MEC) and standard ADxE treatment in course two
  Interventions: Drug: Randomisation course 1 mitoxantrone versus DaunoXome; Drug: Randomisation course 2 ADxE versus FLADx
- Experimental DxEC and standard ADxE (Experimental): Experimental arm with DaunoXome in course one (DxEC) and standard ADxE treatment in course two
  Interventions: Drug: Randomisation course 1 mitoxantrone versus DaunoXome
- Standard arm MEC and experimental FLADx (Experimental): Experimental arm with standard MEC in the first course (MEC) and experimental treatment with FLADx in course two
  Interventions: Drug: Randomisation course 2 ADxE versus FLADx
- Experimental DxEC and experimental FLADx (Experimental): Experimental treatment with DaunoXome in course one (DxEC) and experimental treatment with FLADx in course two
  Interventions: Drug: Randomisation course 1 mitoxantrone versus DaunoXome; Drug: Randomisation course 2 ADxE versus FLADx

INTERVENTIONS:
Drug: Randomisation course 1 mitoxantrone versus DaunoXome — In course one with cytarabine and etoposide either mitoxantrone (standard) or DaunoXome (experimental) is given as anthracycline.
  Arms: Experimental DxEC and experimental FLADx; Experimental DxEC and standard ADxE; Standard arm MEC and ADxE
Drug: Randomisation course 2 ADxE versus FLADx — The second course is randomised to either ADxE (standard arm) or FLADx
  Arms: Experimental DxEC and experimental FLADx; Standard arm MEC and ADxE; Standard arm MEC and experimental FLADx

SUMMARY:
This study evaluates the effect of different induction courses in children and adolescents with newly diagnosed acute myeloid leukemia. In the first course patients are randomised to receive either standard anthracycline therapy with mitoxantrone or experimental DaunoXome. In the second course patients are randomised between standard treatment with ADxE (cytarabine, DaunoXome, etoposide) or experimental therapy with FLADx (fludarabine, cytarabine, DaunoXome).

ELIGIBILITY:
Inclusion Criteria:

1. AML as defined by the WHO diagnostic criteria
2. Age < 19 years at time of diagnosis
3. Written informed consent

Exclusion Criteria:

1. Previous chemotherapy or radiotherapy. This includes patient with secondary AML after previous cancer therapy
2. AML secondary to previous bone marrow failure syndrome.
3. Down syndrome (DS)
4. Acute promyelocytic leukaemia (APL)
5. Myelodysplastic syndrome (MDS)
6. Juvenile Myelomonocytic Leukaemia (JMML)
7. Known intolerance to any of the chemotherapeutic drugs in the protocol.
8. Fanconi anaemia
9. Major organ failure precluding administration of planned chemotherapy.
10. Positive pregnancy test
11. Lactating female or female of childbearing potential not using adequate contraception

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease | On day 22 after the first induction and after second induction
  MRD will be measured by flow cytometry. In the randomisation for course 1 the endpoint is at day 22. In the randomisation for course 2 the endpoint is immediately before start of consolidation

SECONDARY OUTCOMES:
Event-free survival | 5 years
  Event-free survival at five years
Acute toxicity | six months
  Hematological and other organ toxicity after each course
Long-term toxicity | 10 years
  Long-term toxicity in particular cardiac toxicity
Overall survival | Five years
  Overall survival at five years

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Abrahamsson, MD, PhD, Study Chair — Children's Cancer Centre, Queen Silvias Childrens and Adolescents Hospital 416 85 Gothenburg, Sweden; Barbara de Moerloose, MD, PhD, Principal Investigator — Ghent University Hospital, Children´s Hospital, Princess Elisabeth, Department of Pediatric Hematology-Oncology, 3K12D, De Pintelaan 185 - 9000 Gent, Belgium; Ha Shau-Yin, MD, PhD, Principal Investigator — Dept of Paediatrics & Adolescent Medicine, Queen Mary Hospital, The University of Hong Kong, Pokfulam, Hong Kong; Henrik Hasle, MD, PhD, Principal Investigator — Department of Pediatrics, Aarhus University Hospital Skejby 8200 Aarhus N, Denmark; Kirsi Jahnukainen, MD, PhD, Principal Investigator — Division of Hematology-Oncology and Stem Cell Transplantation, Children's Hospital, Helsinki University Central Hospital, PL 281, 00029 Helsinki, Finland; Olafur G Jonsson, MD, PhD, Principal Investigator — Children´s Hospital, Landspitali University Hospital, Hringbraut, 101 Reykjavik, Iceland; Gertjan Kaspers, MD, PhD, Principal Investigator — Department of Pediatrics, VU University Medical Center Amsterdam De Boelelaan 1117, NL-1081 HV Amsterdam, The Netherlands; Birgitte Lausen, MD, PhD, Principal Investigator — Dept of Pediatrics and Adolescent Medicine, Rigshospitalet, University of Copenhagen, Denmark; Josefine Palle, MD, PhD, Principal Investigator — Dept of Woman´s and Children´s Health, Uppsala University, Uppsala, Sweden; Kadri Saks, MD, PhD, Principal Investigator — Tallinn Children's Hospital, Dep. Hematology oncology, Tervise 28, Tallinn 13419, Estonia.; Bernward Zeller, MD, PhD, Principal Investigator — Pediatric Dept, Women and Children's Division, Oslo University Hospital Rikshospitalet, Mailbox 4950 Nydalen, N-0424 Oslo, Norway
Locations (32):
- Belgium (7):
  - HUDERF, L'Hôpital des Enfants Hématologie / Oncologie, Brussels
  - UZ Brussel, Pediatrische Hemato-Oncologie F930, Brussels
  - UCL, Cliniques Universitaires Saint-Luc, Brussels
  - Ghent University Hospital, Children´s Hospital, Princess Elisabeth, Department of Pediatric Hematology-Oncology, Ghent
  - UZ Leuven, Kinder Hemato-Oncologie, Leuven
  - CHR Citadelle, Liège
  - CHC Espérance, Montegnée
- Denmark (2):
  - Department of Pediatrics, Aarhus University Hospital Skejby, Aarhus
  - Dept of Pediatrics and Adolescent Medicine, Rigshospitalet, University of Copenhagen, Copenhagen
- Tallinn Children's Hospital, Dep. Hematology oncology, Tallinn, Estonia
- Finland (5):
  - Division of Hematology-Oncology and Stem Cell Transplantation, Children's Hospital, Helsinki University Central Hospital, Helsinki
  - Department of Pediatrics, Kuopio University Hospital, Kuopio
  - Department of Pediatrics, Oulu University Hospital, Oulu
  - Department of Pediatrics, Tampere University Central Hospital, Tampere
  - Department of Pediatrics, Turku University Central Hospital, Turku
- Dept of Paediatrics & Adolescent Medicine, Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong
- Children´s Hospital, Landspitali University Hospital, Reykjavik, Iceland
- Netherlands (5):
  - VU University Medical Center Department of Pediatric Oncology/Hematology, Amsterdam
  - Emma Children's Hospital/ Amsterdam Medical Center Department of Pediatric Oncology, Amsterdam
  - Department of Pediatric Oncology/Hematology Beatrix childrens hospital / University Medical Center Groningen, Groningen
  - University Medical Center Nijmegen Department of Pediatric Oncology/Hematolog, Nijmegen
  - Erasmus MC - Sophia Childrens Hospital University Medical Center Rotterdam, Rotterdam
- Norway (4):
  - Department of Pediatrics, Haukeland University Hospital, Bergen, Bergen
  - Pediatric Dept, Women and Children's Division, Oslo University Hospital Rikshospitalet, Oslo
  - Department of Pediatrics, University Hospital of North Norway, Tromsoe, Tromsø
  - Department of Cancer and Haemathology, St Olavs Hospital, Trondheim University Hospital, Trondheim
- Sweden (6):
  - Queen Silvias Childrens and Adolescents Hospital, Gothenburg
  - Dept of Pediatrics, Linköpings University Hospital, Linköping
  - Dept of Pediatrics, Skåne University Hospital, Lund
  - Astrid Lindgrens Barnsjukhus, Karolinska University Hospital, Stockholm
  - Dept of Pediatrics, Norrlands University Hospital, Umeå
  - Dept of Pediatrics, Akademiska barnsjukhuset, Uppsala

REFERENCES:
- [Derived] Tierens A, Arad-Cohen N, Cheuk D, De Moerloose B, Fernandez Navarro JM, Hasle H, Jahnukainen K, Juul-Dam KL, Kaspers G, Kovalova Z, Lausen B, Noren-Nystrom U, Palle J, Pasauliene R, Jan Pronk C, Saks K, Zeller B, Abrahamsson J. Mitoxantrone Versus Liposomal Daunorubicin in Induction of Pediatric AML With Risk Stratification Based on Flow Cytometry Measurement of Residual Disease. J Clin Oncol. 2024 Jun 20;42(18):2174-2185. doi: 10.1200/JCO.23.01841. Epub 2024 Apr 11. PMID 38603646